CLINICAL TRIAL: NCT06211946
Title: Comparison of Abdominal Aorta Palpation With Point of Care Ultrasound Imaging Measurements in Healthy Individuals
Brief Title: Abdominal Aorta Palpation With Point of Care Ultrasound Imaging Measurements
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Darren Q. Calley, Principal Investigator, Mayo Clinic
Other Study IDs: 23-009766
Record Dates: First submitted 2024-01-09; First posted 2024-01-18 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Physical Examination; Ultrasound Imaging; Abdominal Aortic Aneurysm
Keywords: Physical Therapy; Abdominal Screening; Ultrasound Imaging
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare the measurements of abdominal aorta width via palpation and point of care ultrasound imaging in healthy individuals. The main question[s] it aims to answer are:

* Is there a measurement difference in abdominal aorta width in healthy individuals as measured by palpation and point of care ultrasound imaging?
* Are palpation measurements and point of care ultrasound imaging measurements reliable when performed by physical therapy researchers? Participants will be asked to have their abdominal area be palpated around the umbilicus and will have ultrasound imaging performed over their abdominal aorta area. It is anticipated participation in the study will take less than 15 minutes. Subjects will be asked to return for a repeat visit within 1 month to determine reliability of measurements.

DETAILED DESCRIPTION:
As part of a review of systems to screen for non-musculoskeletal low back pain, physical therapists perform an abdominal screening exam which may include observation and palpation of the abdominal aorta. Using a two-finger distance palpation method, an estimation of the abdominal aorta width is one screening approach. A growing part of physical therapy practice is use of point of care ultrasound imaging (POCUS) to guide a physical therapy diagnosis and assist with clinical reasoning. No published research could be found on physical therapists using diagnostic ultrasound imaging to measure the abdominal aorta distance, or intra-reliability in palpation of abdominal aorta transverse distance. A measurement in excess of 3 cm is typically characterized as an abdominal aortic aneurism. The goal of this study is to determine the reliability and agreement of abdominal aorta palpation measurements with transverse diameter abdominal aorta POCUS measurements performed by physical therapy researchers in healthy individuals. Healthy patients over the age of 18 without a history of abdominal aortic aneurisms will be recruited for a study with 2 visits within 1 month of each other at Mayo Clinic Rochester. Patients will undergo a brief survey of basic demographic information including age, sex, and race/ethnicity at first visit only. The patients will also have their height and weight taken by the examiners to determine BMI. The order of testing will be randomly allocated. Patients will lie supine in the hook-lying position with the abdomen exposed to the xiphoid process. Study Examiner 1 will take a two-finger palpation measurement of the abdominal aorta, just cranial to the umbilicus and caudal to the xyphoid using a tape measure. For the palpation measurement, the examiner will be blinded to the numerical measurement and another examiner will measure and record the distance. Study Examiner 2 will then perform transverse infra-renal [above the umbilicus and slightly left] abdominal aorta ultrasound using Vscan Air™ ultrasound imaging device. A short axis view of the abdominal aorta will be captured on screen with the borders of the aorta clearly outlined. Using digital calipers, the largest aorta diameter from outer lumen to outer lumen will be measured. Examiner 2 will be blinded to the actual ultrasound measurement, and the measurement will be read and recorded by another examiner. Subjects will return for a follow-up visit to repeat the above process within 1 month to capture intra-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adults > 18 years of age

Exclusion Criteria:

* History of abdominal aortic aneurysm.
* Individuals that are pregnant or trying to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults over the age of 18
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Palpation Measurement | at baseline and within 1 month later
  Palpated width of abdominal aorta will be measured using a tape measure.
Ultrasound Measurement | at baseline and within 1 month later
  Width of abdominal aorta will be measured using point of care ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Calley, P.T., DScPT, OCS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials